CLINICAL TRIAL: NCT00005777
Title: Randomized Trial of Minimal Ventilator Support and Early Corticosteroid Therapy to Increase Survival Without Chronic Lung Disease in Extremely-Low-Birth-Weight Infants
Brief Title: Minimal Breathing Support and Early Steroids to Prevent Chronic Lung Disease in Extremely Premature Infants (SAVE)
Acronym: SAVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was halted because of unanticipated nonrespiratory adverse events related to dexamethasone therapy.
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Waldemar A. Carlo, Lead Principal Investigator, University of Alabama - Birmingham
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0018; U10HD034216 (NIH); U10HD034167 (NIH); U10HD021397 (NIH); U10HD027853 (NIH); U10HD027871 (NIH); U10HD021415 (NIH); U10HD027904 (NIH); U10HD027881 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027880 (NIH); U10HD021373 (NIH); U01HD036790 (NIH); M01RR008084 (NIH); M01RR006022 (NIH); M01RR000750 (NIH); M01RR000997 (NIH); M01RR000070 (NIH); M01RR001032 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Bronchopulmonary Dysplasia; Respiratory Distress Syndrome; Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Chronic Lung Disease (CLD); Dexamethasone; Glucocorticoids; Respiration, Artificial; Mechanical ventilation; Respiratory Insufficiency
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Respiratory Distress Syndrome; Premature Birth; Respiratory Aspiration; Respiratory Insufficiency | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Minimal ventilation with Dexamethasone (Experimental): Minimal ventilator support strategy (permissive hypercapnia) and early stress dose dexamethasone therapy
  Interventions: Procedure: Minimal mechanical ventilation management; Drug: Dexamethasone
- Minimal Ventilation without Dexamethasone (Experimental): Minimal ventilator support strategy (permissive hypercapnia) and no dexamethasone therapy
  Interventions: Procedure: Minimal mechanical ventilation management; Drug: Placebo
- Routine ventilation with Dexamethasone (Active Comparator)
  Interventions: Procedure: Routine mechanical ventilation management; Drug: Dexamethasone
- Routine ventilation without Dexamethasone (Active Comparator)
  Interventions: Procedure: Routine mechanical ventilation management; Drug: Placebo

INTERVENTIONS:
Procedure: Minimal mechanical ventilation management — Partial pressure of carbon dioxide (PCO2) target (>52 mm Hg)
  Arms: Minimal Ventilation without Dexamethasone; Minimal ventilation with Dexamethasone
Procedure: Routine mechanical ventilation management — Partial pressure of carbon dioxide (PCO2) target <48 mm Hg)
  Arms: Routine ventilation with Dexamethasone; Routine ventilation without Dexamethasone
Drug: Dexamethasone — Treatment with the study medication was initiated within 24 hours after birth. The dexamethasone-treated infants received a 10-day tapered course (0.15 mg of dexamethasone per kilogram per day for three days, followed by 0.10 mg per kilogram for three days, 0.05 mg per kilogram for two days, and 0.02 mg per kilogram for two days), with the daily dose divided in half and given at 12-hour intervals intravenously or orally, if an intravenous catheter was no longer in place.
  Arms: Minimal ventilation with Dexamethasone; Routine ventilation with Dexamethasone
Drug: Placebo — The infants in the placebo groups received equal volumes of saline.
  Other Names: Saline
  Arms: Minimal Ventilation without Dexamethasone; Routine ventilation without Dexamethasone

SUMMARY:
This multicenter clinical trial tested whether minimal ventilation decreases death or BPD. Infants with birth weight 501g to 1000g and mechanically ventilated before 12 hours were randomly assigned to minimal ventilation (partial pressure of carbon dioxide [PCO(2)] target >52 mm Hg) or routine ventilation (PCO(2) target <48 mm Hg) and a tapered dexamethasone course or saline placebo for 10 days, using a 2 x 2 factorial design. The primary outcome was death or BPD at 36 weeks' postmenstrual age. Blood gases, ventilator settings, and FiO2 were recorded for 10 days; complications and outcomes were monitored to discharge. The infants' neurodevelopment was evaluated at 18-22 months corrected age.

DETAILED DESCRIPTION:
Chronic lung disease (CLD), also known as bronchopulmonary dysplasia (BPD), in very premature infants has been associated with mechanical ventilation and relative adrenal insufficiency.

This multicenter clinical trial tested whether minimal ventilation decreases death or BPD. Infants with birth weight 501g to 1000g and mechanically ventilated before 12 hours were randomly assigned to minimal ventilation (partial pressure of carbon dioxide [PCO(2)] target >52 mm Hg) or routine ventilation (PCO(2) target <48 mm Hg) and a tapered dexamethasone course or saline placebo for 10 days, using a 2 x 2 factorial design. The primary outcome was death or BPD at 36 weeks' postmenstrual age. Blood gases, ventilator settings, and FiO2 were recorded for 10 days; complications and outcomes were monitored to discharge.

The trial was terminated by the Steering Committee when the interim analysis for the Data Safety and Monitoring Committee showed a higher rate of spontaneous gastrointestinal perforations in the dexamethasone-treated infants.

Neurodevelopment was assessed at 18-22 months postmenstrual age.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 12 hrs of age and less than 10 days chronologic age
* 501-1000 gm
* Intubated and mechanically ventilated before 12 hrs
* Indwelling vascular catheter
* Infants 751-100 gm must be receiving FiO2 greater than 0.30 and have received at least 1 dose of surfactant at randomization
* Parental consent

Exclusion Criteria:

* Major congenital anomaly
* Symptomatic non-bacterial infection
* Permanent neuromuscular conditions that affect respiration
* Terminal illness (defined as pH values less than 6.8 for more than 2 hours or persistent bradycardia associated with hypoxia for more than 2 hours)
* Use of postnatal corticosteroids

Ages: 5 Minutes to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 1998-02; Primary Completion 1998-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Death or moderate to severe bronchopulmonary dysplasia | 36 weeks postmenstrual age

SECONDARY OUTCOMES:
Death | 36 weeks postmenstrual age
Mechanical ventilation | 36 weeks postmenstrual age
Pulmonary interstitial emphysema | 36 weeks postmenstrual age
Pneumothorax | 36 weeks postmenstrual age
Open-label steroids | 36 weeks postmenstrual age
Reintubation | 36 weeks postmenstrual age
Intracranial hemorrhage (IVH) III or IV | 36 weeks postmenstrual age
Periventricular leukomalacia | 36 weeks postmenstrual age
Necrotizing enterocolitis | 36 weeks postmenstrual age
Duration of oxygen supplementation | 36 weeks postmenstrual age
Duration of ventilation | 36 weeks postmenstrual age
Length of hospitalization | Hospital discharge
Death or neurodevelopmental impairment | 18-22 months corrected age
Death | 18-22 months corrected age
Neurodevelopmental impairment | 18-22 months corrected age
Cerebral palsy | 18-22 months corrected age
Bilateral blindness | 18-22 months corrected age
Deafness | 18-22 months corrected age
Bayley Scales of Infant Development-Revised II Psychomotor Developmental Index (PDI) | 18-22 months corrected age
Rehospitalizations | 18-22 months corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A. Carlo, MD, Study Director — University of Alabama at Birmingham; Ann R. Stark, MD, Study Director — Brigham and Women's Hospital; William Oh, MD, Principal Investigator — Brown University, Women & Infants Hospital; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies & Children's Hospital; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Barbara J. Stoll, MD, Principal Investigator — Emory University; Charles R. Bauer, MD, Principal Investigator — University of Miami; Lu-Ann Papile, MD, Study Director — University of New Mexico; David K. Stevenson, MD, Principal Investigator — Stanford University; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Jon E. Tyson, MD MPH, Principal Investigator — University of Texas Southwestern Medical Center; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; W. Kenneth Poole, PhD, Principal Investigator — RTI International
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - RTI International, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Result] Carlo WA, Stark AR, Wright LL, Tyson JE, Papile LA, Shankaran S, Donovan EF, Oh W, Bauer CR, Saha S, Poole WK, Stoll B. Minimal ventilation to prevent bronchopulmonary dysplasia in extremely-low-birth-weight infants. J Pediatr. 2002 Sep;141(3):370-4. doi: 10.1067/mpd.2002.127507. PMID 12219057
- [Result] Stark AR, Carlo WA, Tyson JE, Papile LA, Wright LL, Shankaran S, Donovan EF, Oh W, Bauer CR, Saha S, Poole WK, Stoll BJ; National Institute of Child Health and Human Development Neonatal Research Network. Adverse effects of early dexamethasone treatment in extremely-low-birth-weight infants. National Institute of Child Health and Human Development Neonatal Research Network. N Engl J Med. 2001 Jan 11;344(2):95-101. doi: 10.1056/NEJM200101113440203. PMID 11150359
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org